CLINICAL TRIAL: NCT05882994
Title: The Effect of Range of Motion Exercises on Fatigue and Sleep Quality in Hemodialysis Patients: Randomized Controlled Study
Brief Title: The Effect of Range of Motion Exercises on Fatigue and Sleep Quality in Hemodialysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, İLKNUR ÖRS, Director, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Necmettin Erbakan Üniversty
Record Dates: First submitted 2023-05-08; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Renal Failure
Keywords: Renal Failure; Exercises; Fatigue; Sleep quality
MeSH Terms: conditions — Renal Insufficiency; Motor Activity; Fatigue; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: After obtaining the consent of 44 patients who met the inclusion criteria of the study, the selection of the patients to form the sample will be made at random according to the patient list in which the patient names in the institution are determined in alphabetical order and numbers. Two groups will be formed with at least one patient in each group, using a simple randomization method created on a computer (www.randomizer.org) by an independent researcher who was not involved in the study.
Who Masked: Outcomes Assessor
Masking Description: single
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rom exercise (Experimental): In this study, ROM exercises will be applied by the researcher 2 days a week for 12 weeks to the intervention group separated by simple randomization method.In this study, considering the existing literature, it was planned to apply the exercise to the patients twice a week, for 12 weeks, with 5 minutes of warm-up, 15 minutes of rom exercises , and 5 minutes of cooling down . Range of motion exercises include wrist rotation (clockwise and counterclockwise), wrist flexion and extension. elbow joint full flexion and extension; rotating ankles (clockwise and counterclockwise); and full flexion and extension of the ankles will be performed. Each movement will be made 20 rounds per minute. The researcher will have the patients perform rom exercises and supervise them during the exercise .
  Interventions: Behavioral: rom exercise
- control group (No Intervention): Patients in the control group will receive routine care during hemodialysis.At the beginning of the study, participants will be asked to fill out data collection tools consisting of Personal Information Form, Piper Fatigue Scale, Pittsburgh Sleep Quality Index. Data will be collected with data collection tools in the 6th and 12th weeks.

INTERVENTIONS:
Behavioral: rom exercise — At the beginning of the study, participants will be asked to fill out data collection tools consisting of Personal Information Form, Piper Fatigue Scale, Pittsburgh Sleep Quality Index. Data will be collected with data collection tools in the 6th and 12th weeks. Evaluation will be done. At the end of the study, rom exercises will be applied to the patients in the control group.
  Arms: rom exercise

SUMMARY:
Range of motion exercises is a simple nursing action that has many benefits and is easy to perform independently . Hemodialysis patients are less active and have low intrinsic motivation for physical activity compared to sedentary healthy individuals. The aim of this study is to determine the effect of joint range of motion exercises on fatigue and sleep quality in patients receiving hemodialysis treatment. As a result of the literature review; The lack of a study on this subject and the inclusion of nurses, who play an important role in symptom management, in care interventions that are easy to learn and without complications, increase the quality of care.

DETAILED DESCRIPTION:
In the advanced stage of chronic kidney disease, hemodialysis treatment is required to maintain the well-being of patients and improve their quality of life.It has been reported in the literature that the prevalence of fatigue varies between 60-97% in patients undergoing hemodialysis . Fatigue is a subjective feeling of weakness, loss of energy, tiredness and weakness. As a result of fatigue, patients experience limited participation in life and feel dependent. They often experience failure to be understood by others and meet expectations. This affects patients' self-esteem and causes problems with changing roles and relationships, identity, and meaning in life.

One of the most common complaints due to various reasons in patients receiving hemodialysis treatment is deterioration in sleep quality. In different studies conducted in patients receiving hemodialysis treatment, it has been reported that the deterioration in sleep quality varies between 53.3% and 87% . Deterioration in sleep quality, on the other hand, causes a decrease in patients' daily life activities, energy levels, self-care power and quality of life .

The quality of life has improved significantly, especially in the symptoms and effects of kidney disease. Range of another method of reducing the level of fatigue, is an activity or physical exercise to keep the body healthy, improve health, and maintain physical health. Range of motion is good for increasing cardiac output, alveolar ventilation, basal metabolic rate and joint mobilization. It is also a good option for reducing weakness and increasing stress tolerance.

Nurses have responsibilities in the symptom management of HD treatment, which reduces the quality of life of the patients, increases the stress level and negatively affects the physical and psychosocial aspects, supports the patients better, increases their quality of life, and provides evidence. Hemodialysis patients are inactive for an average of 12 hours per week during hemodialysis. By adding more functionality to the time spent on hemodialysis, it can improve patients' quality of life and increase compliance with treatment. The aim of this study is to determine the effect of range of motion exercises on the fatigue and sleep quality experienced by patients receiving hemodialysis treatment. As a result of the literature review, it was necessary to carry out this study in order not to carry out a study on this subject and to include nurses who play an important role in symptom management in their care interventions, which are easy to learn and do not have any complications, and to improve the quality of care with their applications. The aim of the study is to determine the effect of range of motion exercises applied to hemodialysis patients on fatigue and sleep quality.

METHOD: It was designed as a parallel group randomized controlled study. Reporting of the study will adhere to the CONSORT scheme for parallel group randomized trials.

Management:In the current hemodialysis unit, patients receive hemodialysis treatment in bed. In the study, ROM application will be applied on the same day of hemodialysis treatment. In the literature, it is recommended to apply exercise for 15 minutes in the first 2 hours of the hemodialysis session. Since patients experience fluid accumulation in the body before hemodialysis begins, such excess fluids should be removed within 4-5 hours. This rapid release of fluids from the body can sometimes lead to hemodynamic changes and symptoms such as hypotension or cramping. Because Based on the literature review recommendations of specialist physicians and nurses, the best time for intervention will be considered 30 minutes after the start of dialysis and during the first 2 hours of dialysis .

In this study, considering the existing literature, it was planned to apply range of motion exercises to patients twice a week, for 12 weeks and for 15 minutes. Range of motion exercises include wrist rotation (clockwise and counterclockwise), wrist flexion and extension. elbow joint full flexion and extension; rotating ankles (clockwise and counterclockwise); and full flexion and extension of the ankles will be performed. Each movement will be made 20 rounds per minute. The co-investigator will have the intervention group undergo ROM and supervise them during hemodialysis. The investigator will pay attention to the comfort of the patients and whether they experience problems such as shortness of breath, fatigue or nausea during the intervention .

Before ROM exercises, the patients in the intervention group will be checked for blood pressure and pulse.

Control group patients will be given routine treatment and care. After the research is completed, ROM exercises will be performed on the control group.

Application:

When the implementation phase of the research begins, the purpose of the research will be explained and written/verbal consent will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years,

  * literate,
  * Receiving hemodialysis treatment for at least 6 months,
  * Hemodialysis patients who volunteered to participate in the study will be included in the study.

Exclusion Criteria:

* Having an additional disease that triggers fatigue (advanced COPD, heart failure, asthma, cancer, etc.),

  * Hearing and communication problems,
  * Having a psychiatric diagnosis (major depression etc.),
  * History of myocardial infarction or unstable angina in the last 12 months
  * Severe uncontrolled diabetes
  * Uncontrolled hypertension with systolic blood pressure >200 mmHg and/or diastolic blood pressure >120 mmHg,
  * Those with tendon, ligament or muscle tear, Unhealed fracture,
  * Patients with deep vein thrombosis will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-06-15 (Estimated); Primary Completion 2023-10-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Piper Fatigue Scale | 6 weeks after the first assessment
  The behavioral sub-dimension consists of six items, the affective sub-dimension consists of five items, the sensory sub-dimension consists of five items, and the cognitive sub-dimension consists of six items. Sub-dimension scores and total fatigue score are calculated over a total of 22 items. In the calculation of the total fatigue score, all scores of 22 items are added and divided by the number of items. 0 points obtained as a result of the average score; you have no fatigue, 1-3 points are "light tiredness", 4-6 points are "moderate tiredness", 7-10.
Pittsburgh Sleep Quality Index (PUKI) | 6 weeks after the first assessment
  PUKI is an index that evaluates sleep quality in the last month and consists of 19 questions and 7 components. The total score has a value between 0-21, a high total score indicates poor sleep quality. A total PSQI score of ≤5 means "good sleep" and >5 means "bad sleep".

CONTACTS AND LOCATIONS:
Overall Officials: Selda Arslan, Study Director — Selda Arslan, Phd Study Director Necmettin Erbakan University Faculty of Nursing; ilknur örs, Principal Investigator — Study Principal İnvestigator

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Effect of Intradialytic Range of Motion Exercise on Dialysis Adequacy and Fatigue in Hemodialysis Patients — https://pubmed.ncbi.nlm.nih.gov/35767683/
- See also: The effect of intradialytic aerobic exercise on dialysis efficacy in hemodialysis patients: a randomized controlled trial — https://pubmed.ncbi.nlm.nih.gov/35767683/